CLINICAL TRIAL: NCT01532388
Title: Randomized Controlled Trial of eScreen for Problematic Drug Use
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Anne H Berman, Affiliated Researcher, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2008/308-31/5D
Record Dates: First submitted 2011-10-27; First posted 2012-02-14 (Estimated); Results first posted 2020-09-29 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Problematic AOD Use
Keywords: Randomized Controlled Trial; Alcohol; Drugs; Internet; Screening; Brief intervention

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- eScreen (Experimental): Web based self-monitoring of problematic alcohol and drug use.
  Interventions: Behavioral: eScreen
- Control group (No Intervention): Untreated control group

INTERVENTIONS:
Behavioral: eScreen — Web based self-monitoring of problematic alcohol and drug use.
  Arms: eScreen

SUMMARY:
Objectives: This study compared the efficacy of eScreen in a two-armed randomized controlled design, measuring outcomes in terms of changes in problematic drug use up to one year after study recruitment. The eScreen brief Internet intervention for problematic alcohol and drug use offers self-screening, in-depth self-reporting, personalized feedback and treatment recommendations as well as an electronic diary. Progress over time is shown in diagrams detailing consumption levels.

Method: Participants with only problematic drug use according to the Drug Use Disorders Identification Test (DUDIT),(DUDIT >0 for both men and women) or both problematic alcohol use according to the Alcohol Use Disorders Identification Test (AUDIT), (AUDIT >7 for men and AUDIT >5 for women) and drug use were randomized to T1 (n=101) or the control group (n=101). Outcomes on alcohol and/or drug use as well as health-related symptoms were assessed after 3, 6 and 12 months.

Hypotheses that were tested in this study are 1) that both groups would reduce their drug consumption and drug-related problems at follow-ups compared to the baseline level and 2) that participants in the eScreen group would reduce their drug consumption and drug-related problems to a higher extent than participants in the control group (no intervention) at follow-ups.

DETAILED DESCRIPTION:
Background: The aim of this study is to investigate the effects of an Internet-based screening and brief intervention (SBI) site for problematic alcohol and drug use among illicit drug users.

Method: Individuals searching for information about alcohol or drugs online who scored over 0 on the Drug Use Disorders Identiﬁcation Test (DUDIT) and were 15 years or older were recruited for this trial and randomized into one group receiving Internet-based screening and brief intervention via eScreen.se(n = 101) or one assessment-only control group (n = 101). Both groups were screened at baseline and followed up at 3 and 6 months. The primary outcome measure was the DUDIT-C score and secondary outcome measures were DUDIT, AUDIT-C (Alcohol Use Disorders Identiﬁcation Test-C) and AUDIT scores.Additional outcomes included the proportion of drug abstainers and those who made a clinically signiﬁcant change in their alcohol and drug use. Four statistical models of analysis were used to conservatively assess results.

ELIGIBILITY:
Inclusion Criteria:

* DUDIT >0

Exclusion Criteria:

* DUDIT = 0

Ages: 15 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 202 (Actual)
Dates: Start 2009-09; Primary Completion 2011-04 (Actual); Study Completion 2012-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Anne H Berman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet, Department of Clinical Neurosciene, Stockholm, Sweden

REFERENCES:
- [Background] Sinadinovic K, Berman AH, Hasson D, Wennberg P. Internet-based assessment and self-monitoring of problematic alcohol and drug use. Addict Behav. 2010 May;35(5):464-70. doi: 10.1016/j.addbeh.2009.12.021. Epub 2010 Jan 4. PMID 20092953
- [Background] Sinadinovic K, Wennberg P, Berman AH. Population screening of risky alcohol and drug use via Internet and Interactive Voice Response (IVR): a feasibility and psychometric study in a random sample. Drug Alcohol Depend. 2011 Mar 1;114(1):55-60. doi: 10.1016/j.drugalcdep.2010.09.004. Epub 2010 Oct 27. PMID 21030164
- [Result] Sinadinovic K, Wennberg P, Berman AH. Targeting problematic users of illicit drugs with Internet-based screening and brief intervention: a randomized controlled trial. Drug Alcohol Depend. 2012 Nov 1;126(1-2):42-50. doi: 10.1016/j.drugalcdep.2012.04.016. Epub 2012 May 20. PMID 22613182
- [Result] Sinadinovic K, Wennberg P, Berman AH. Internet-based screening and brief intervention for illicit drug users: a randomized controlled trial with 12-month follow-up. J Stud Alcohol Drugs. 2014 Mar;75(2):313-8. doi: 10.15288/jsad.2014.75.313. PMID 24650825
- See also: Anne H Berman's profile at Uppsala University — https://www.katalog.uu.se/profile/?id=N19-2760
- See also: Web based self-monitoring site — https://escreen.se/Default.aspx?ReturnUrl=%2f

RESULTS

PARTICIPANT FLOW:
Period: 3-month Follow-up
Arm/Group | eScreen | Control Group
Started | 101 | 101
Completed | 33 | 33
Not Completed | 68 | 68
Not completed — Lost to Follow-up | 68 | 68
Period: 6-month Follow-up
Arm/Group | eScreen | Control Group
Started | 101 (All participants registered in the trial were contacted for follow-ups at 3, 6 and 12 months.) | 101 (All participants registered in the trial were contacted for follow-ups at 3, 6 and 12 months.)
Completed | 27 | 35
Not Completed | 74 | 66
Not completed — Lost to Follow-up | 74 | 66
Period: 12-month Follow-up
Arm/Group | eScreen | Control Group
Started | 101 (All participants registered in the trial were contacted for follow-ups at 3, 6 and 12 months.) | 101 (All participants registered in the trial were contacted for follow-ups at 3, 6 and 12 months.)
Completed | 32 | 34
Not Completed | 69 | 67
Not completed — Lost to Follow-up | 69 | 67

BASELINE CHARACTERISTICS:
Population: All individuals who have registered for the study and registered mandatory baseline data have been included in the baseline analyses.
Groups:
- Total: Total of all reporting groups
Arm/Group | eScreen | Control Group | Total
Number analyzed (Participants) | 101 | 101 | 202
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 5 | 4 | 9
  Between 18 and 65 years | 95 | 95 | 190
  >=65 years | 1 | 2 | 3
Age, Continuous [Mean (Standard Deviation); unit: years] | 33.16 (13.34) | 31.93 (12.37) | 32.54 (12.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 48 | 42 | 90
  Male | 53 | 59 | 112
Region of Enrollment [Number; unit: participants]
  Sweden | 101 | 101 | 202

OUTCOME MEASURES:

1. Primary Outcome: Drug Use Disorders Identification Test-Consumption (DUDIT-C)
Description: The primary outcome measure for this trial was the total DUDIT score for the first four DUDIT questions at 3-month follow-up, as a measure of drug consumption only, referred to as the DUDIT-C.The DUDIT-C is a measure including the first four items of the DUDIT, with a minimum score of 0 and a maximum score of 16. Higher scores mean a worse outcome. Regarding the DUDIT-C, you will find information on it in the following articles. Please note that the analyses all refer to the same sample from a randomized controlled trial. Apart from the data in the two articles describing results from the current study, there are additional analyses shown in:
  Berman, A. H., Wennberg, P., & Sinadinovic, K. (2015). Changes in Mental and Physical Well-Being Among Problematic Alcohol and Drug Users in 12-Month Internet-Based Intervention Trials. Psychology of Addictive Behaviors, 29(1), 97-105. doi: 10.1037/a0038420 A higher score means a worse outcome.
Time Frame: 3 months
Population: The analyses have been carried out according to both the Intention To Treat method (ITT) and according to Per protocols method (PP).
  Where possible, missing values were imputed with last observation carried backwards. In cases where no follow-up data were available, the last observation was carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 4.8 (3.9) | 4.5 (4.1)

2. Secondary Outcome: Drug Use Disorders Identification Test (DUDIT)
Description: The total DUDIT score at 3-month follow-up, as a summarized measure of drug use (including drug consumption and drug-related problems). The DUDIT, an 11-item scale, has a minimum score of 0 and a maximum score of 44. Higher scores mean a worse outcome.
Time Frame: 3 months
Population: The analyzes have been carried out according to both the Intention To Treat method (ITT) and according to Per protocols method (PP).
  Where possible, missing values were imputed with last observation carried backwards. In cases where no follow-up data were available, the last observation was carried forward.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 12.0 (12.6) | 10.6 (12.1)

3. Secondary Outcome: Alcohol Use Disorders Identification Test - Consumption (AUDIT-C)
Description: The total AUDIT score for the first three AUDIT questions at 3-month follow-up, as a measure of alcohol consumption only, referred to as the AUDIT-C. The AUDIT-C, a 3-item scale, has a minimum score of 0 and a maximum score of 12. Higher scores mean a worse outcome.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 6.9 (3.1) | 6.7 (3.4)

4. Secondary Outcome: Alcohol Use Disorders Identification Test - AUDIT
Description: The total AUDIT score at 3-month follow-up, as a summarized measure of alcohol use (including alcohol consumption and alcohol-related problems). The AUDIT, an 10-item scale, has a minimum score of 0 and a maximum score of 40. Higher scores mean a worse outcome.
Time Frame: 3 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 18.5 (10.1) | 17.7 (10.9)

5. Secondary Outcome: Drug Use Disorders Identification Test-Consumption (DUDIT-C)
Description: The total DUDIT score for the first four DUDIT questions at 6-month follow-up, as a measure of drug consumption only, referred to as the DUDIT-C.The DUDIT-C is a measure including the first four items of the DUDIT, with a minimum score of 0 and a maximum score of 16. Higher scores mean a worse outcome.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 4.7 (4.2) | 4.2 (4.1)

6. Secondary Outcome: Drug Use Disorders Identification Test (DUDIT)
Description: The total DUDIT score at 6-month follow-up, as a summarized measure of drug use (including drug consumption and drug-related problems). The DUDIT, an 11-item scale, has a minimum score of 0 and a maximum score of 44. Higher scores mean a worse outcome.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 11.6 (12.8) | 10.4 (12.2)

7. Secondary Outcome: Alcohol Use Disorders Identification Test-Consumption (AUDIT-C)
Description: The total AUDIT score for the first three AUDIT questions at 6-month follow-up, as a measure of alcohol consumption only, referred to as the AUDIT-C. The AUDIT-C, a 3-item scale, has a minimum score of 0 and a maximum score of 12. Higher scores mean a worse outcome.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 6.5 (3.3) | 6.5 (3.4)

8. Secondary Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: The total AUDIT score at 6-month follow-up, as a summarized measure of drug use (including alcohol consumption and alcohol-related problems). The AUDIT, an 10-item scale, has a minimum score of 0 and a maximum score of 40. Higher scores mean a worse outcome.
Time Frame: 6 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 17.4 (10.7) | 17.3 (10.7)

9. Secondary Outcome: Drug Use Disorders Identification Test-Consumption (DUDIT-C)
Description: The total DUDIT score for the first four DUDIT questions at 12-month follow-up, as a measure of drug consumption only, referred to as the DUDIT-C.The DUDIT-C is a measure including the first four items of the DUDIT, with a minimum score of 0 and a maximum score of 16. Higher scores mean a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 4.4 (4.2) | 4.0 (4.1)

10. Secondary Outcome: Drug Use Disorders Identification Test (DUDIT)
Description: The total DUDIT score at 12-month follow-up, as a summarized measure of drug use (including drug consumption and drug-related problems). The DUDIT, an 11-item scale, has a minimum score of 0 and a maximum score of 44. Higher scores mean a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 11.0 (12.8) | 9.9 (12.2)

11. Secondary Outcome: Alcohol Use Disorders Identification Test-Consumption (AUDIT-C)
Description: The total AUDIT score for the first three AUDIT questions at 12-month follow-up, as a measure of alcohol consumption only, referred to as the AUDIT-C. The AUDIT-C, a 3-item scale, has a minimum score of 0 and a maximum score of 12. Higher scores mean a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 6.3 (3.3) | 6.5 (3.4)

12. Secondary Outcome: Alcohol Use Disorders Identification Test (AUDIT)
Description: The total AUDIT score at 12-month follow-up, as a summarized measure of drug use (including alcohol consumption and alcohol-related problems). The AUDIT, an 10-item scale, has a minimum score of 0 and a maximum score of 40. Higher scores mean a worse outcome.
Time Frame: 12 months
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | eScreen | Control Group
Number analyzed (Participants) | 101 | 101
units on a scale | 16.9 (10.8) | 17.1 (10.5)

ADVERSE EVENTS:
Time Frame: 13 months from baseline recruitment.
Arm/Group | eScreen | Control Group
Serious Adverse Events (participants affected / at risk) | 0/101 | 0/101
Other Adverse Events (participants affected / at risk) | 0/101 | 0/101

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No